CLINICAL TRIAL: NCT07257562
Title: A Prospective Observational Study on the Effects of Concomitant Administration of Bacteroides Fragilis and Branched-Chain Amino Acids on HBsAg Clearance
Brief Title: Combined Use of Bacteroides Fragilis and BCAAs on HBsAg Clearance
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MRCTA, ECFAH of FMU [2023]082
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PegIFNα2b+Nucleoside analog: The patients receive both PegIFNα2b and Nucleoside analog therapy.
  Interventions: Drug: PegIFNα2b+Nucleoside analog
- PegIFNα2b+Nucleoside analog+Bacteroides fragilis+Branched-Chain Amino Acids: The patients received the concomitant administration of Bacteroides fragilis and Branched-Chain Amino Acids, supplemented to their ongoing combination therapy with PegIFNα2b and Nucleoside analog.
  Interventions: Drug: PegIFNα2b+Nucleoside analog+Bacteroides fragilis+Branched-Chain Amino Acids

INTERVENTIONS:
Drug: PegIFNα2b+Nucleoside analog — The patients receive both PegIFNα2b and Nucleoside analog therapy.
  Groups: PegIFNα2b+Nucleoside analog
Drug: PegIFNα2b+Nucleoside analog+Bacteroides fragilis+Branched-Chain Amino Acids — The patients received the concomitant administration of Bacteroides fragilis and BCAA, supplemented to their ongoing combination therapy with PegIFNα2b and Nucleoside analog.
  Groups: PegIFNα2b+Nucleoside analog+Bacteroides fragilis+Branched-Chain Amino Acids

SUMMARY:
The goal of this prospective observational study is to determine the effects of concomitant administration of Bacteroides fragilis and Branched-Chain Amino Acids on hepatitis B virus clearance. The primary question it aims to answer is whether this concomitant administration can promote HBV clearance.

The study will observe the HBV clearance rate in chronic hepatitis B patients who receive Bacteroides fragilis and BCAA as a supplement to their routine antiviral therapy. For comparison, researchers will compare the clearance rate in this group to that observed in a control group of chronic hepatitis B patients receiving a standard antiviral regimen based on PegIFNα2b and nucleoside analogs.

ELIGIBILITY:
Inclusion Criteria:

- chronic hepatitis B patients

Exclusion Criteria:

* patients with malignancies
* patients with other liver diseases
* pregnancy patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with chronic hepatitis B who are receiving both PegIFNα2b and nucleoside analog therapy with or without concomitant administration of Bacteroides fragilis and Branched-Chain Amino Acids.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
HBsAg clearance | 48 months
  HBsAg clearance is confirmed when two consecutive measurements, taken at an interval of at least 2 weeks, demonstrate HBsAg levels below the assay's lower limit of detection (< 0.05 IU/mL) as quantitatively determined by the Abbott Architect-i2000SR system with Chemiluminescent Microparticle Immunoassay (CMIA) technology.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
The goal of this prospective observational study is to determine the effects of concomitant administration of Bacteroides fragilis and Branched-Chain Amino Acids on hepatitis B virus clearance. The primary question it aims to answer is whether this concomitant administration can promote HBV clearance.
  The study will observe the HBV clearance rate in chronic hepatitis B patients who receive Bacteroides fragilis and BCAA as a supplement to their routine antiviral therapy. For comparison, researchers will compare the clearance rate in this group to that observed in a control group of CHB patients receiving a standard antiviral regimen based on PegIFNα2b and nucleoside analog.
Supporting Information: Study Protocol